CLINICAL TRIAL: NCT00311636
Title: Prevention of Chemotherapy-induced Menopause by Temporary Ovarian Suppression With Triptorelin Vs. Control in Young Breast Cancer Patients. A Randomized Phase III Multicenter Study [PROMISE]
Brief Title: Triptorelin in Preventing Early Menopause in Premenopausal Women Who Are Receiving Chemotherapy for Stage I, Stage II, or Stage III Breast Cancer That Has Been Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Mammella (GIM) (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: GIM-6; CDR0000468839 (Registry Identifier: PDQ (Physician Data Query)); GIM-PROMISE; EU-20606; GIM-5104
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2008-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; Epirubicin; Fluorouracil; Methotrexate; Paclitaxel; Triptorelin Pamoate; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Drug: paclitaxel
Drug: triptorelin
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Chemotherapy may cause early menopause in premenopausal women. Triptorelin may prevent this from happening.

PURPOSE: This randomized phase III trial is studying triptorelin to see how well it works in preventing early menopause in premenopausal women who are receiving chemotherapy for stage I, stage II, or stage III breast cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the incidence of chemotherapy-induced early menopause in premenopausal women undergoing adjuvant chemotherapy in combination with vs without triptorelin for previously resected stage I-III breast cancer.

Secondary

* Compare the toxicity of adjuvant chemotherapy and triptorelin vs adjuvant chemotherapy alone.

OUTLINE: This is a prospective, open-label, multicenter, randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (adjuvant chemotherapy alone): Patients receive adjuvant chemotherapy alone.
* Arm II (adjuvant chemotherapy and triptorelin): Patients receive adjuvant chemotherapy and triptorelin intramuscularly 1 week before and then every 4 weeks for the duration of chemotherapy. The last dose of triptorelin is given before the last course of chemotherapy.

Patients with hormone-sensitive tumors who resume ovarian function after stopping chemotherapy and triptorelin restart triptorelin until ovarian function is suppressed for 2 years.

Patients undergo menopausal status assessment, using follicle-stimulating hormone, luteinizing hormone, and estradiol as biochemical markers, at baseline and 3, 6, 9, and 12 months after the last course of chemotherapy.

After completion of study treatment, patients are followed at 3, 6, 9, and 12 months.

PROJECTED ACCRUAL: A total of 280 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer resected at time of original diagnosis

  * Stage I-III disease
* Candidate for 1 of the following adjuvant chemotherapy regimens:

  * FEC (fluorouracil, epirubicin hydrochloride, and cyclophosphamide) every 21 or 28 days
  * CMF (cyclophosphamide, methotrexate, and fluorouracil) every 28 days
  * A→CMF (doxorubicin hydrochloride followed by CMF)
  * EC→P (epirubicin hydrochloride and cyclophosphamide every 21 days followed by paclitaxel every 21 days)
  * FEC→P (FEC every 21 days followed by paclitaxel every 21 days)
  * EC→D (EC every 21 days followed by docetaxel every 21 days)
  * AC (doxorubicin hydrochloride and cyclophosphamide) every 21 days
  * AC→P (AC every 21 days followed by paclitaxel every 21 days)
  * E→CMF (epirubicin hydrochloride followed by CMF every 28 days)
* No evidence of metastases or localized or distant recurrence

  * Investigation to exclude metastases required for any suspicious manifestation
* Premenopausal, defined as the presence of active menstrual cycles or normal menses within six weeks before initiation of chemotherapy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or adequately treated in situ carcinoma of the cervix
* No history of noncompliance to medical regimens or patients who are considered potentially unreliable
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy and/or radiotherapy for cancer or non-neoplastic disease
* No other concurrent hormonal therapy except for tamoxifen

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2003-09; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-induced early menopause as measured by follicle-stimulating hormone, 17 beta estradiol levels, and menstrual activity resumption at 1 year following the completion of chemotherapy

SECONDARY OUTCOMES:
Toxicity as measured by Common Toxicity Criteria at each chemotherapy course

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Del Mastro, MD, Study Chair — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (18):
- Italy (18):
  - Ospedale Civile, Castelfranco - TV
  - Ospedale Sant Anna, Como
  - Ospedale Santa Croce, Cuneo
  - Azienda Ospedaliera di Firenze, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Presidio Ospedaliero di Livorno, Livorno
  - Carlo Poma Hospital, Mantova
  - Federico II University Medical School, Naples
  - Seconda Universita di Napoli, Naples
  - Istituto G. Pascale, Naples
  - Ospedale Silvestrini, Perugia
  - Ospedale Santa Chiara Pisa, Pisa
  - Istituto Regina Elena, Rome
  - Ospedale Civile ASL 1, Sassari
  - Ospedale SS Trinita, Sora
  - Ospedale Treviglio Caravaggio, Treviglio
  - Ospedale Maggiore dell' Universita, Trieste
  - Universita di Torino, Turin

REFERENCES:
- [Result] Del Mastro L, Boni L, Michelotti A, Gamucci T, Olmeo N, Gori S, Giordano M, Garrone O, Pronzato P, Bighin C, Levaggi A, Giraudi S, Cresti N, Magnolfi E, Scotto T, Vecchio C, Venturini M. Effect of the gonadotropin-releasing hormone analogue triptorelin on the occurrence of chemotherapy-induced early menopause in premenopausal women with breast cancer: a randomized trial. JAMA. 2011 Jul 20;306(3):269-76. doi: 10.1001/jama.2011.991. PMID 21771987
- [Derived] Lambertini M, Boni L, Michelotti A, Gamucci T, Scotto T, Gori S, Giordano M, Garrone O, Levaggi A, Poggio F, Giraudi S, Bighin C, Vecchio C, Sertoli MR, Pronzato P, Del Mastro L; GIM Study Group. Ovarian Suppression With Triptorelin During Adjuvant Breast Cancer Chemotherapy and Long-term Ovarian Function, Pregnancies, and Disease-Free Survival: A Randomized Clinical Trial. JAMA. 2015 Dec 22-29;314(24):2632-40. doi: 10.1001/jama.2015.17291. PMID 26720025